CLINICAL TRIAL: NCT06711783
Title: VISAN - Vårdkedja I Samverkan För Unga Patienter Med Anorexia Nervosa (collaborative Chain of Care in Adolescnt Anorexia Nervosa Treatment)
Brief Title: Treatment of Adolescent Anorexia Nervosa
Acronym: VISAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 281931
Record Dates: First submitted 2024-11-25; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Eating Disorders
Keywords: anorexia nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Family based treatment (Experimental): Family based treatment including the whole chain of care, such as day care and in patiant care when necessary. The interventions includes consultation with dietician, psyciotherapist, LEAP-Y and Skills training based on an individual plan.
  Interventions: Behavioral: Family based therapy

INTERVENTIONS:
Behavioral: Family based therapy — Family based therapy following the Maudsley model

SUMMARY:
VISAN is a naturalistic study of family based treatment of Anorexia nervosa in adolescnet girls.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with f500 or f501 and being planned for family based therapy at the unit.

Exclusion Criteria:

* being subjected to care by the social welfare system

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Remission | End of treatment (assessed up to 1 year)
  No longer fulfilling criteria for an eating disorder

CONTACTS AND LOCATIONS:
Locations (1):
- Orebro eating disorder unit, Örebro, Örebro County, Sweden